CLINICAL TRIAL: NCT00003580
Title: Phase II Study - Efficacy of Amifostine in Alleviating Toxicity Associated With Targeted Supradose Cisplatin and Concomitant Radiation Therapy (RADPLAT) in Head and Neck Cancer
Brief Title: Amifostine to Treat Side Effects of Treatment in Patients Receiving Radiation Therapy and Cisplatin for Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Tennessee (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: UTENN-6507; CDR0000066647 (Registry Identifier: PDQ (Physician Data Query)); ALZA-98-066-ii; NCI-V98-1472
Record Dates: First submitted 1999-11-01; First posted 2004-05-25 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2006-05

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Head and Neck Cancer; Oral Complications; Radiation Toxicity
Keywords: oral complications; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; drug/agent toxicity by tissue/organ; radiation toxicity
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Head and Neck Neoplasms; Radiation Injuries; Squamous Cell Carcinoma of Head and Neck | interventions — Amifostine; Cisplatin; Radiotherapy

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: cisplatin
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Drugs such as amifostine may protect normal cells from the side effects of chemotherapy and radiation therapy.

PURPOSE: Phase II trial to study the effectiveness of amifostine in treating side effects of treatment in patients receiving radiation therapy and cisplatin for advanced head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of amifostine in alleviating treatment related mucositis associated with targeted supradose cisplatin and concurrent radiotherapy (RADPLAT protocol) in patients with stage III or IV squamous cell carcinoma of the head and neck. II. Determine the efficacy of amifostine in alleviating other treatment related morbidities associated with this protocol in these patients.

OUTLINE: This is an open label, multicenter study of amifostine. Patients receive external beam radiotherapy 5 days a week for approximately 6.5-7.5 weeks. Concurrent with radiotherapy, patients receive amifostine IV over 10 minutes, 30 minutes prior to cisplatin, then cisplatin intra-arterially over 3-5 minutes. Chemotherapy and amifostine course is repeated every week for 4 weeks. Patients are followed at 1 month.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued into this study over 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed squamous cell carcinoma of the oral cavity, nasopharynx, oropharynx, hypopharynx, or larynx Previously untreated Stage III or IV No distant metastatic disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hepatic: SGOT and SGPT no greater than 2.5 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL Creatinine clearance greater than 61 mL/min Other: No history of any underlying medical or psychiatric illness Not pregnant or nursing Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: No prior therapy for head and neck cancer Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: At least 24 hours since prior antihypertensive medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-06; Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K. Thomas Robbins, MD, Study Chair — University of Florida
Locations (1):
- William F. Bowld Hospital, Memphis, Tennessee, United States